CLINICAL TRIAL: NCT06512727
Title: Testing the Pain Relief of musculOskeletal Conditions and Arthritis Using Culturally Tailored InterVentions for Black Elders (PROACTIVE) Intervention: A Randomized Controlled Trial
Brief Title: The PROACTIVE Study for Black Elders
Acronym: PROACTIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB202302085; 1R01NR021183-01 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Pain; Chronic Pain; Osteoarthritis; Pain, Chronic; Movement Evoked Pain
Keywords: chronic musculoskeletal pain; chronic pain; Black; African Americans; pain self-management; prayer; social determinants of health
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Control Group) (No Intervention): The control group will continue their usual pain treatment and self-management (SM) routines.
  Participations will not receive in-depth culturally congruent education, prayer skills, or financial counseling. Usual care is expected to vary between participants.
- PROACTIVE (Experimental): This is a four-session pain self-management (SM) intervention designed to reduce movement-evoked pain by providing participants with behavioral support that addresses social determinants of health: (1) culturally congruent SM education + SM resource toolkit, (3) active prayer support, and (3) financial counseling.
  Interventions: Behavioral: PROACTIVE Intervention

INTERVENTIONS:
Behavioral: PROACTIVE Intervention — Duration: Once-weekly face-to-face sessions Session Time: 1.5-2 hours Intervention: (1) culturally congruent self-management (SM) education and + SM resource toolkit, (3) active prayer support, and (3) financial counseling/insurance navigation Reinforcement: daily ecological momentary intervention support using Apple smartwatches
  Other Names: FAITH (Finding Arthritis Interventions That Help)
  Arms: PROACTIVE

SUMMARY:
Chronic musculoskeletal pain (CMP), while a leading cause of physical disablement, is a neglected national health disparity issue in Black communities. The purpose of this study is to test a novel culturally congruent pain self-management intervention. A total of 120 persons aged 50-92, self-identifying as Black or African American having CMP will be invited to participate in this study. The primary outcome measured throughout this 3-year study is movement-evoked pain (MEP).

DETAILED DESCRIPTION:
Chronic musculoskeletal conditions and their primary source of pain, movement-evoked pain (MEP), causes significant pain interference, long-term mobility impairment, healthcare costs, and psychosocial inequalities. MEP affects more Black/African Americans (B/AAs) and is reported as more severe than in White participants. Compounded by race, age, and more disadvantageous social determinants of health (SDoH), this unequal burden of pain becomes even greater in health disparity populations like older B/AAs. Many B/AA older adults rely on non-pharmacological pain self-management (SM) strategies. Yet, current chronic musculoskeletal pain (CMP) SM interventions do not measure MEP as a primary endpoint nor address faith/spirituality, Black culture, and other underlying potentially modifiable SDoH (e.g., health literacy, financial hardship). The investigator team propose to enhance older B/AAs' capacity to manage MEP by investigating the effects of a socioculturally congruent pain SM intervention (Pain Relief for musculOskeletal conditions and Arthritis using Culturally-Tailored InterVentions for Black Elders [PROACTIVE]). This intervention will provide culturally congruent pain SM education with a SM resource toolkit, active prayer skills, and financial counseling to explain participants' healthcare/insurance benefits for pain care. This study will enroll 120 B/AAs (50 years and older) with CMP into a parallel group, single-blind, randomized controlled trial to test whether PROACTIVE decreases MEP in the immediate post-intervention period (n= 60) (Aim 1) and over time (Sub-Aim 1a) compared to a usual care control group (n= 60). To determine efficacy, this study will use state-of-the-art and real-time technologies to measure primary outcome as well as pain interference, pain coping, and physical function (secondary outcomes) (Sub-Aim 1b). The PROACTIVE group will work with a faith-community nurse and financial counselor over four weeks to enhance knowledge of CMP SM, utilization of active prayer and faith, and financial literacy of health insurance benefits and resources available to cover treatments for pain. Each weekly session will last up to 2 hours and will be followed by six days of ecological momentary assessments of pain and SM outcomes and ecological momentary interventions guiding participants through weekly SM practice skills. A fourth booster session will reinforce content and training and help sustain SM. Another goal is to examine the differential effects of PROACTIVE on MEP according to demographic (sex as a biological variable, gender, age), psychosocial, and SDoH factors (Aim 2). The proposed intervention is expected to produce meaningful reductions in MEP in B/AA older adults experiencing disabling chronic musculoskeletal conditions. Ideally, this study will identify precision behavior targets and responders to inform intervention refinement. This study is innovative because it: (1) addresses three key social determinants of health central to B/AAs' pain experience- health literacy, faith, and finances, (2) embeds community-engaged research methodologies, (3) tests active prayer as a novel faith-based, culturally relevant intervention, (4) uses real-time ecological momentary assessment (EMA) to measure pain and related outcomes and use just-in-time ecological momentary interventions (EMI) to deliver pain SM decision support and active prayers, and (5) measures MEP as a primary endpoint in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as being part of the Black American diaspora (Black/African American, Afro-Caribbean)
2. Age 50-92 years
3. Self-report chronic musculoskeletal pain (CMP) as defined as persistent or recurrent pain lasting 6 months or longer that arises as part of a disease or injurious process directly affecting bone(s), joint(s), muscle(s), or related soft tissue(s)
4. Self-report a chronic musculoskeletal condition (e.g., osteoarthritis, chronic low back pain) in at least one lower extremity joint (hip, knee, low back, or ankle pain)
5. Report chronic musculoskeletal symptoms: aching, stiffness, or swelling in a major lower extremity joint or low back on most days (4-5/7) of the week
6. Have (or be eligible for) a healthcare insurance plan in the state of Florida (Medicare, Medicaid, Medicare Advantage plans, Blue Cross/Blue Shield, Humana, Aetna, etc.)
7. Able to read, write, and understand English at sixth-grade level

Exclusion Criteria:

1. Unwilling to be randomized to either study arm
2. Self-reported diagnosis of sickle cell disease or related thalassemias
3. History of major neurological event (e.g., stroke) or current neurological disease (e.g., Parkinson's disease, multiple sclerosis, epilepsy)
4. Major cardiovascular problem in the past 6 months that would cause shortness of breath and/or chest pain (e.g. myocardial infarction, coronary artery bypass graft, or valve replacement, pulmonary embolism or deep venous thrombosis) or uncontrolled Hypertension (Systolic Blood Pressure (SBP) > 170 mmHg, Diastolic Blood Pressure (DBP) > 90 mmHg) OR Hypotension (SBP <90 mmHg, DBP <60 mmHg)
5. Currently undergoing curative or palliative chemotherapy or radiation for active cancer
6. Severe physical impairment (e.g., a major activity of daily living disability requiring use of wheelchair as primary method of mobility, or unable to dress, bath, use the toilet, or transfer independently)
7. Serious mental health disorder requiring hospitalization within past 12 months
8. Severe sensory deficit (severe hearing loss or blindness)

Ages: 50 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in movement-evoked pain from baseline to 4 weeks (post-intervention) | Baseline, Week 4, 1-month, 3-months
  Defense and Veterans Pain Rating Scale (DVPRS) is a validated, self-reported and preferred pain scale for assessing pain intensity and its impact on activities. Possible scores range from 0 (no pain) to 10 (as bad as it could be). Movement-evoked pain (MEP) intensity during the Short Physical Performance Battery (SPPB), a physical performance test that evaluates lower extremity functioning by assessing: standing balancing, gait speed, and repeated chair stand ability.
  Change:
  1. Week 4 score - Baseline score
  2. 1 month score - Baseline score
  3. 3-months score - Baseline score

SECONDARY OUTCOMES:
Pain interference | Baseline, Week 4, 1-month, 3-months
  PROMIS (Patient-Reported Outcomes Measurement Information System) Adult Short Form v1.0- Pain interference 6b, a is a validated, 6-item self-report instrument with strong reliability and validity. Pain interference measures the degree of interference with usual social, work, physical, and emotional functioning. Questions ask people to recall how much pain has interfered social, cognitive, emotional, physical, and recreational activities in the last seven day (1=not at all to 5=very much).
Pain coping | Baseline, Week 4, 1-month, 3-months
  Coping Strategies Questionnaire is a valid and reliable survey with six cognitive (diverting attention, reinterpreting pain sensations, coping self-statements, ignoring pain sensations, praying or hoping, and catastrophizing) and one behavioral (increasing activity level) pain coping subscales where 0 (never do) to 6 (always do that when in pain). A score from 0-36 points is calculated for each subscale.
Physical function- Short Physical Performance Battery | Baseline, Week 4, 1-month, 3-months
  Performance-based activities, such as the Short Physical Performance Battery (SPPB) will evaluate physical function. The SPPB measures standing balance, 4-meter gait speed, and ability to rise from chair. Each task is score 0-4 and total scores range from 0-12, with lower scores indicating greater impairment.
Physical function- 3-Minute Walk | Baseline, Week 4, 1-month, 3-months
  The 3-minute walk test requires participants to walk continuously for 3 minutes, and it measures endurance and aerobic capacity. Time walked, number of meters walked, and pain intensity (i.e., MEP) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Staja Q Booker, PhD, RN, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Public Use Data: All deidentified study data that are not designated as restricted use will be made available as public use data to the research community. Users of public data must agree to terms of use from Mendeley Data repository and the PI, which are designed to protect study participants. Data users also agree not to share or redistribute any data downloads. The dataset can only be used for studying health or biomedical conditions.
  Restricted Access Data: Data that are determined to be potentially identifiable through indirect or deductive disclosure are provided under restricted data contract to users who demonstrate a valid research need and meet conditions of use. These restricted data will include separate files with geospatial indicators below the level of state, such as county, census tract, block-group, and block for all years; and linkages to contextual social determinants of health data.
Supporting Information: SAP
Time Frame: After the study is complete, the study team will submit all remaining scientific data to the data repository and will update the randomized controlled trial status to "complete" in clinicaltrials.gov. Scientific data will be made available to other users approximately 12 months following the final data collection point or within the award period (or NCE) if requested, and remain available for an indefinite time or for as long as it is scientifically useful for the research community, institutions, and/or the broader public.
Access Criteria: Researchers requesting data directly from the PI will need to complete a "Data Sharing and Use Agreement" prior to release of data. The requesting institution's Institutional Review Board or equivalent body must approve the requested use or provide documentation of exemption before data will be shared.